CLINICAL TRIAL: NCT02900040
Title: The French DIVAT: a Clinical Database Associated With a Biological Banking Accessible to Initiate Epidemiological and Translational Collaborative Researches in Kidney Transplantation
Brief Title: Clinical Database Associated With a Biological Banking Accessible to Initiate Epidemiological and Translational Collaborative Researches in Kidney Transplantation
Acronym: DIVAT
Status: Recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC12_0452
Record Dates: First submitted 2016-09-09; First posted 2016-09-14 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Kidney Transplantation
MeSH Terms: interventions — Kidney Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Years
Biospecimen Retention: Samples With DNA — peripheral blood cells, serum, plasma, urine, m-RNA, and DNA of recipients and donors
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- patients with kidney transplantations: patients with kidney transplantations
  Interventions: Other: kidney transplantation

INTERVENTIONS:
Other: kidney transplantation

SUMMARY:
The French DIVAT (standing for Données Informatisées et VAlidées en Transplantation in french, and in English "Computerized and VAlidated Data in Transplantation" ) cohort was Kicked off in 1994 by the Transplantation Urology Nephrology Institute of the Nantes University Hospital in France. The primary objective of this multicenter computerized database was to enable prospective clinical and epidemiological research studies concerning kidney transplant recipients, particularly focusing on mid- and long-term clinical outcomes, therapeutic strategies and public health issues. The patient-case system of the DIVAT cohort allows the monitoring of medical records of all patient-specific and allograft-specific data, including bio-banking since 2005. Data are collected from the date of transplantation until the graft failure, at each scheduled outpatient visit or hospital admission motivating by a new clinical, therapeutical or biological expression. The DIVAT cohort contains information on more than 11000 transplant recipients between 1994 and today, issued from 8 French university hospitals centers (the DIVAT Network is organized by a consortium agreement). 18% of all patients underwent retransplantation and 11% of all kidney transplants originated from living donors. The DIVAT network heavily works to ensure a high-quality data collection with the aim of exploring adequately the complex post-transplantation process. The Divat network encourage collaborations and enables interested researchers to submit a research project by completing a request form available on the DIVAT website (http://www.divat.fr/en) describing the context, objectives and design of the study

ELIGIBILITY:
Inclusion Criteria:

* over the age of 18 years
* with renal transplant

Exclusion Criteria:

* minor
* pediatric transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eight French transplantation centers participate to the DIVAT network: Nantes, Paris Necker, Nancy and Montpellier since 1994, Toulouse since 1997, Lyon since 2006, and Paris Saint-Louis and Nice that joined the network since 2013. All patients over the age of 18 years, who received a renal transplant, are included. No other particular inclusion criteria exist.
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 1994-01; Primary Completion 2050-01 (Estimated); Study Completion 2050-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with Overall Survival | 2 years
Proportion of participants with Overall Survival | 4 years
Proportion of participants with Overall Survival | 6 years

SECONDARY OUTCOMES:
expansion of effector memory CD8+ T cells dosage | 1 year
  potential marker for acute graft dysfunction
expansion of effector memory CD8+ T cells dosage | 6 years
  potential marker for late graft dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: Magali Giral, PU-PH, Principal Investigator — Nantes Universuty Hospital
Locations (8):
- France (8):
  - Docteur Buron, Lyon
  - Professeur Mourad, Montpellier
  - Professeur Kessler, Nancy
  - Professeur Ladriere, Nancy
  - Pr Cassuto, Nice
  - Professeur Kreis, Paris
  - Professeur Legendre, Paris
  - Professeur Rostaing, Toulouse

REFERENCES:
- [Derived] Choisy C, Foucher Y, Masset C, Maanaoui M, Lenain R, Rostaing L, Jouve T, Le Quintrec M, Serre JE, Morelon E, Charmetant X, Ladriere M, Girerd S, Sicard A, Gosset C, Mariat C, Claisse G, Giral M, Dantan E; DIVAT Consortium. Identification of Donor-recipient Interactions for a Relative Appraisal of Kidney Graft Marginality: A French Multicentric Cohort-based Study. Transplantation. 2025 Dec 1;109(12):e708-e717. doi: 10.1097/TP.0000000000005464. Epub 2025 Jul 14. PMID 40653616
- [Derived] Danger R, Le Berre L, Cadoux M, Kerleau C, Papuchon E, Mai HL, Nguyen TV, Guerif P, Morelon E, Thaunat O, Legendre C, Anglicheau D, Lefaucheur C, Couzi L, Del Bello A, Kamar N, Le Quintrec M, Goutaudier V, Renaudin K, Giral M, Brouard S; DIVAT Consortium. Subclinical rejection-free diagnostic after kidney transplantation using blood gene expression. Kidney Int. 2023 Jun;103(6):1167-1179. doi: 10.1016/j.kint.2023.03.019. Epub 2023 Mar 27. PMID 36990211